CLINICAL TRIAL: NCT02285439
Title: Phase I-II Study of MEK 162 for Children With Low-Grade Gliomas and Other Ras/Raf/ERK Pathway Activated Tumors
Brief Title: Study of MEK162 for Children With Low-Grade Gliomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Nathan Robison, M.D., Medical Director of Inpatient Services, Attending Neuro-Oncologist, Associate Professor, Children's Hospital Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-15-00146
Record Dates: First submitted 2014-10-09; First posted 2014-11-07 (Estimated); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Low-Grade Gliomas; Malignant Neoplasms, Brain; Soft Tissue Neoplasms
Keywords: Pediatric Oncology; Ras/Raf pathway; Low-Grade Glioma; MEK inhibitor
MeSH Terms: conditions — Brain Neoplasms; Soft Tissue Neoplasms | interventions — binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 (Experimental): Patients with non-hematologic malignancies that are recurrent, progressive, or refractory after standard up-front therapy receiving MEK162 will define the MTD, DLT, and toxicity profile.
  Interventions: Drug: MEK162
- Phase 2 (Experimental): Children with recurrent tumors signaling through the Ras/Raf pathway will be treated in 3 strata to define the activity of MEK162. S1: Children with LGG characterized by a BRAF truncated fusion (KIAA1549 and similar translocations). S2: Children with NF1 and LGG. S 3: Children with tumors involving the Ras/Raf pathway not included in strata 1 or 2.
  Interventions: Drug: MEK162
- Target Validation (Experimental): Patients eligible for phase 2 (any stratum) for whom tumor biopsy or resection is clinically indicated may be enrolled on the target validation arm. Patients will receive MEK162 for 7 to 21 days prior to their surgery. Tumor sample will be analyzed for drug concentration and target inhibition.
  Interventions: Drug: MEK162

INTERVENTIONS:
Drug: MEK162 — • MEK162 is currently supplied as film-coated tablets in dose strength of 15 mg. The film-coated tablets consist of MEK162 drug substance, lactose monohydrate, microcrystalline cellulose, colloidal silicon dioxide, croscarmellose sodium, magnesium stearate, and a commercial film coating. The original tablets are yellow to dark yellow capsule-shaped
  Other Names: ARRY 438162; Binimetinib

SUMMARY:
The goal of this clinical trial is to study the drug MEK162 in children with a brain tumor call low-grade glioma, as well as in children with other tumors in which a specific growth signal is abnormally turned on. The main questions it aims to answer are:

What is the correct dose of MEK162 in children? What are the side effects of MEK162 in children? Is MEK162 effective in children with low-grade glioma?

Participants on the study receive MEK162 by mouth twice daily for up to 2 years.

DETAILED DESCRIPTION:
PROTOCOL SUMMARY:

Phase 1: Patients with non-hematologic malignancies that are recurrent, progressive, or refractory after standard up-front therapy receiving MEK162 will define the maximum tolerated dose (MTD), dose-limiting toxicities (DLT), and toxicity profile.

Phase 2: Patients with recurrent or progressive tumors signaling through the ras/raf pathway after standard up-front therapy will be treated in three strata to define the activity of MEK162.

Stratum 1: Pediatric patients with recurrent or progressive low-grade glioma (LGG) characterized by a BRAF truncated fusion (KIAA1549 and similar translocations).

Stratum 2: Pediatric patients with neurofibromatosis type 1 (NF1) and recurrent or progressive LGG.

Stratum 3: Pediatric patients with recurrent or progressive tumors thought to involve the ras/raf/MAP pathway but not included in strata 1 or 2. This includes any LGG not included in strata 1 or 2 (i.e., any LGG without a BRAF truncated fusion in a patient without NF1), any tumor other than LGG in a patient with NF1, and any other tumor with a known activating BRAF, NRAS or KRAS mutation.

Target validation phase: Patient enrolled on the phase 2 component (any stratum) for whom tumor biopsy or resection is clinically indicated. Patients will receive MEK162 for 7 to 21 days prior to their surgery. Samples will be analyzed for concentration of drug and target inhibition.

Length of therapy:

Protocol treatment will last approximately 48 weeks from the start of MEK162 in the absence of significant toxicity. Treatment will be administered based on the dose escalation schema for phase 1. Patients in the phase 2 component of the trial will also receive a planned 48 weeks of therapy. Those undergoing planned tumor resection based on clinical criteria will be eligible to receive 7-21 days of treatment with MEK162 prior to the surgical procedure.

Imaging to assess response will be obtained at the end of cycle 1 (+/- 1 week), at the end of cycle 3 (+/- 2 weeks) and after every three cycles thereafter (+/- 2 weeks). A cycle will consist of 28 days (+/- 3 days) and MEK162 will be given continuously. Patients deriving benefit may continue therapy beyond study completion but all protocol specific evaluations (other than survival or progression) will conclude after one year. All patients will be followed with progression as the end point.

ELIGIBILITY:
Patients with recurrent or progressive disease, as defined in the following three strata below, will be eligible. For eligibility determination, tumor imaging from at least two time-points must be available to document radiographic progression or recurrence. Patients with non-progressive refractory tumors will not be eligible.

* Stratum 1: patients with LGG with a BRAF truncated fusion that is measurable in at least two dimensions on imaging.
* Stratum 2: patients with NF1 and LGG that is measurable in at least two dimensions on imaging.
* Stratum 3: Pediatric patients with a recurrent or progressive tumor thought to involve the Ras/Raf/ERK pathway but not included in strata 1 or 2 that is measurable in at least two dimensions on imaging. This includes any LGG not included in strata 1 or 2 (i.e., any LGG without a BRAF truncated fusion in a patient without NF1), any tumor other than LGG in a patient with NF1, and any other tumor with a documented activating BRAF, NRAS, or KRAS mutation.
* Stratum 4 (surgical arm, target validation): Patients who meet criteria for stratum 1, 2, or 3 for whom tumor biopsy and/or resection is clinically indicated.
* Tumor tissue for correlative studies must be available for all patients except those with NF1 and LGG (stratum 2) or any patient with optic pathway glioma (stratum 2 or 3), for whom tumor tissue is optional.
* Patients must have received at least one prior chemotherapy or radiation regimen prior to progression.
* At the time of enrollment, at least 6 weeks must have elapsed since the last dose of any nitrosourea, and the longer of 2 weeks or 3 half-lives must have elapsed since the last dose of any other tumor-directed medication. or biologic therapy.
* At least 3 months must have elapsed since the last dose of irradiation to the target tumor(s) at the time of enrollment.
* Patients must be >1 year and <18 years old.
* Performance Score using the Karnofsky Performance Scale (patients > 12 years old) or Lansky Play - Performance Scale (patients ≤ 12 years old) must be ≥ 60 assessed within two weeks prior to enrollment.
* Participants must have normal organ and marrow function as defined below within two weeks prior to enrollment:

  * Absolute neutrophil count > 1,000/mcL
  * Platelets > 75,000/mcL and > 7 days since last platelet transfusion. Hemoglobin > 9 gm/dL and > 7 days since last red blood cell transfusion
  * Not refractory to red cell or platelet transfusions
  * Hepatic: Total bilirubin ≤ 1.5 times the upper limit of normal; SGPT (ALT) and SGOT (AST) < 3 times the institutional upper limit of normal
  * Renal: Serum creatinine which is less than 1.5 time the upper limit of institutional normal for age or GFR > 70 ml/min/1.73m2
  * QTc interval < 450ms
  * Left ventricular ejection fraction (LVEF) > 50% as determined by an echocardiogram
* Female patients of childbearing potential must have negative serum or urine pregnancy test within 72 hours of the first dose of MEK162. Patient must not be pregnant or breast-feeding. Patients of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study and for 30 days following cessation of treatment.
* Patient must be able to take oral/enteral medication.
* Patient, parent, or legal guardian must be able to understand and willing to provide informed consent.
* Patients must have recovered from the effects of prior therapy.

Exclusion Criteria

Patients with any of the following characteristics will not be eligible:

* Patients for whom other curative or established standard-of-care therapeutic options with acceptable morbidity exist.
* Patients with any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.
* History of Gilbert's syndrome
* Patients receiving any other anticancer or experimental drug therapy.
* Use of hematopoietic growth factors within 2 weeks prior to initiation of therapy.
* Any other investigational agents within 2 weeks or ≤ 3 half-lives (whichever is longer) before start of study therapy.
* Patients who have undergone surgery ≤ 3 weeks or who have not recovered from side effects of this procedure prior to receiving study drug.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, impaired gastrointestinal function, or psychiatric illness/social situations that would limit compliance with study requirements.
* History or current evidence of retinal vein occlusion (RVO) or predisposing factors to RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes).
* History of retinal degenerative disease
* Prior therapy with a MEK inhibitor
* Impairment of gastrointestinal function (e.g., active ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome)
* Patients who have a neuromuscular disorder that is associated with elevated CK (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
* Patients with uncontrolled hypertension

Inclusion of Women, Minorities, and Other Underrepresented Populations This protocol is open to males and females of all races. See Inclusion Criteria above regarding specific eligibility requirements for female and male patients of child-bearing or child-fathering potential, respectively.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2025-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Robison, MD, Principal Investigator — CHLA
Locations (15):
- United States (15):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Heath Systems, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospitals and Clinics of Minnesota-Minneapolis, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - New York University, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - University of Texas Southwestern Medical, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Dose Level 1: Starting dose of 16 mg/m2/dose BID (twice a day) for patients with recurrent, refractory, or progressive non-hematologic malignancies (CNS or solid tumors) associated with activation of the RAS/RAF/ERK pathway, including any low grade glioma (LGG), any tumor in a patient with NF1, or any tumor with a documented activating BRAF, NRAS, or KRAS mutation, will be eligible. LGG is defined as any WHO grade I or II (or equivalent) astrocytic, oligodendroglial, and/or glioneuronal tumor.
- Phase I Dose Level 2: Starting dose of 20 mg/m2/dose BID (twice a day) for patients with recurrent, refractory, or progressive non-hematologic malignancies (CNS or solid tumors) associated with activation of the RAS/RAF/ERK pathway, including any low grade glioma (LGG), any tumor in a patient with NF1, or any tumor with a documented activating BRAF, NRAS, or KRAS mutation, will be eligible. LGG is defined as any WHO grade I or II (or equivalent) astrocytic, oligodendroglial, and/or glioneuronal tumor.
- Phase I Dose Level 3: Starting dose of 24 mg/m2/dose BID (twice a day) for patients with recurrent, refractory, or progressive non-hematologic malignancies (CNS or solid tumors) associated with activation of the RAS/RAF/ERK pathway, including any low grade glioma (LGG), any tumor in a patient with NF1, or any tumor with a documented activating BRAF, NRAS, or KRAS mutation, will be eligible. LGG is defined as any WHO grade I or II (or equivalent) astrocytic, oligodendroglial, and/or glioneuronal tumor.
- Phase I Dose Level 4: Starting dose of 28 mg/m2/dose BID (twice a day) for patients with recurrent, refractory, or progressive non-hematologic malignancies (CNS or solid tumors) associated with activation of the RAS/RAF/ERK pathway, including any low grade glioma (LGG), any tumor in a patient with NF1, or any tumor with a documented activating BRAF, NRAS, or KRAS mutation, will be eligible. LGG is defined as any WHO grade I or II (or equivalent) astrocytic, oligodendroglial, and/or glioneuronal tumor.
- Phase I Dose Level 5: Starting dose of 32 mg/m2/dose BID (twice a day) for patients with recurrent, refractory, or progressive non-hematologic malignancies (CNS or solid tumors) associated with activation of the RAS/RAF/ERK pathway, including any low grade glioma (LGG), any tumor in a patient with NF1, or any tumor with a documented activating BRAF, NRAS, or KRAS mutation, will be eligible. LGG is defined as any WHO grade I or II (or equivalent) astrocytic, oligodendroglial, and/or glioneuronal tumor.
- Phase II Stratum 1: Starting dose of 32 mg/m2/dose BID (twice a day) for patients with a recurrent or progressive low grade glioma (LGG) with a BRAF truncated fusion that is measurable in at least two dimensions on imaging
- Phase II Stratum 2: Starting dose of 32 mg/m2/dose BID (twice a day) for NF1 patients with a recurrent or progressive low grade glioma (LGG) that is measurable in at least two dimensions on imaging
- Phase II Stratum 3: Starting dose of 32 mg/m2/dose BID (twice a day) for patients with a recurrent or progressive tumor thought to involve the Ras/Raf/ERK pathway but not included in Stratum 1 or 2. This includes any low grade glioma (LGG) not included in Stratum 1 or 2 (any LGG without a BRAF truncated fusion in a patient without NF1), any tumor other than LGG in a patient with NF1, and any other tumor with a documented activating BRAF, NRAS, or KRAS mutation.
- Phase II Stratum 4 - Surgical Arm, Target Validation: Starting dose of 32 mg/m2/dose BID (twice a day) continuous administration for 7-21 days followed by biopsy or resection. Then restarting BID administration after surgery. For patients who meet criteria for stratum 1, 2, or 3 for whom tumor biopsy and/or resection is clinically indicated. Re-institute MEK162 BID after recovery from tumor resection.
Period: Overall Study
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level 2 | Phase I Dose Level 3 | Phase I Dose Level 4 | Phase I Dose Level 5 | Phase II Stratum 1 | Phase II Stratum 2 | Phase II Stratum 3 | Phase II Stratum 4 - Surgical Arm, Target Validation
Started | 4 | 3 | 3 | 3 | 6 | 27 | 22 | 30 | 7
Dose Limiting Toxicity Evaluable (Patients were evaluable for dose limiting toxicity (DLT) if they had a DLT in Cycle 1 or had ≥ 85% of Cycle 1 doses) | 3 | 3 | 3 | 3 | 6 | 26 | 20 | 28 | 7
Completed (Completed defined as completing at least the first 12 cycles of therapy) | 3 | 2 | 3 | 0 | 3 | 9 | 17 | 23 | 5
Not Completed | 1 | 1 | 0 | 3 | 3 | 18 | 5 | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Phase I Dose Level 1: Starting dose of 16 mg/m2/dose BID for patients with recurrent, refractory, or progressive non-hematologic malignancies (CNS or solid tumors) associated with activation of the RAS/RAF/ERK pathway, including any LGG, any tumor in a patient with NF1, or any tumor with a documented activating BRAF, NRAS, or KRAS mutation, will be eligible. LGG is defined as any WHO grade I or II (or equivalent) astrocytic, oligodendroglial, and/or glioneuronal tumor.
- Phase I Dose Level 2: Starting dose of 20 mg/m2/dose BID for patients with recurrent, refractory, or progressive non-hematologic malignancies (CNS or solid tumors) associated with activation of the RAS/RAF/ERK pathway, including any LGG, any tumor in a patient with NF1, or any tumor with a documented activating BRAF, NRAS, or KRAS mutation, will be eligible. LGG is defined as any WHO grade I or II (or equivalent) astrocytic, oligodendroglial, and/or glioneuronal tumor.
- Phase I Dose Level 3: Starting dose of 24 mg/m2/dose BID for patients with recurrent, refractory, or progressive non-hematologic malignancies (CNS or solid tumors) associated with activation of the RAS/RAF/ERK pathway, including any LGG, any tumor in a patient with NF1, or any tumor with a documented activating BRAF, NRAS, or KRAS mutation, will be eligible. LGG is defined as any WHO grade I or II (or equivalent) astrocytic, oligodendroglial, and/or glioneuronal tumor.
- Phase I Dose Level 4: Starting dose of 28 mg/m2/dose BID for patients with recurrent, refractory, or progressive non-hematologic malignancies (CNS or solid tumors) associated with activation of the RAS/RAF/ERK pathway, including any LGG, any tumor in a patient with NF1, or any tumor with a documented activating BRAF, NRAS, or KRAS mutation, will be eligible. LGG is defined as any WHO grade I or II (or equivalent) astrocytic, oligodendroglial, and/or glioneuronal tumor.
- Phase I Dose Level 5: Starting dose of 32 mg/m2/dose BID for patients with recurrent, refractory, or progressive non-hematologic malignancies (CNS or solid tumors) associated with activation of the RAS/RAF/ERK pathway, including any LGG, any tumor in a patient with NF1, or any tumor with a documented activating BRAF, NRAS, or KRAS mutation, will be eligible. LGG is defined as any WHO grade I or II (or equivalent) astrocytic, oligodendroglial, and/or glioneuronal tumor.
- Phase II Stratum 1: Starting dose of 32 mg/m2/dose BID for patients with a recurrent or progressive LGG with a BRAF truncated fusion that is measurable in at least two dimensions on imaging
- Phase II Stratum 2: Starting dose of 32 mg/m2/dose BID for NF1 patients with a recurrent or progressive LGG that is measurable in at least two dimensions on imaging
- Phase II Stratum 3: Starting dose of 32 mg/m2/dose BID for patients with a recurrent or progressive tumor thought to involve the Ras/Raf/ERK pathway but not included in stratum 1 or 2 that is measurable in at least two dimensions on imaging. This includes any LGG not included in strata 1 or 2 (i.e., any LGG without a BRAF truncated fusion in a patient without NF1), any tumor other than LGG in a patient with NF1, and any other tumor with a documented activating BRAF, NRAS, or KRAS mutation.
- Phase II Stratum 4 (Surgical Arm, Target Validation: Starting dose of 32 mg/m2/dose BID for patients who meet criteria for stratum 1, 2, or 3 for whom tumor biopsy and/or resection is clinically indicated.
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level 2 | Phase I Dose Level 3 | Phase I Dose Level 4 | Phase I Dose Level 5 | Phase II Stratum 1 | Phase II Stratum 2 | Phase II Stratum 3 | Phase II Stratum 4 (Surgical Arm, Target Validation | Total
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 6 | 27 | 22 | 30 | 7 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 3 | 3 | 3 | 6 | 27 | 22 | 30 | 7 | 105
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 1 | 3 | 14 | 12 | 13 | 4 | 55
  Male | 2 | 0 | 0 | 2 | 3 | 13 | 10 | 17 | 3 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 1 | 2 | 2 | 7 | 0 | 14
  Not Hispanic or Latino | 3 | 3 | 2 | 1 | 5 | 24 | 19 | 22 | 6 | 85
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 3 | 2 | 11
  White | 3 | 2 | 3 | 1 | 4 | 21 | 19 | 20 | 3 | 76
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 2 | 1 | 3 | 2 | 5 | 2 | 16

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (Strata 1 and 2)
Description: For each stratum, the percentage of patients achieving at least a minor response (defined as greater than or equal to 25% decrease in maximal two dimensional measurements compared to baseline) during the first 12 cycles (nominally 48 weeks) of treatment will be reported.
Time Frame: 48 weeks
Population: Phase II Stratum 2 population n=22; Analysis population n=21. One patient enrolled to this stratum did not initiate treatment and was excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Stratum 1 | Phase II Stratum 2
Number analyzed (Participants) | 27 | 21
Participants | 15 | 12

2. Primary Outcome: 12 Cycle Progression-free and Overall Survival (Strata 1 and 2)
Description: Progression free and overall survival will be reported as Kaplan-Meier estimate who are alive without disease progression, alive with disease progression, deceased without disease progression, and deceased with disease progression 12 cycles (48 weeks) after treatment initiation.
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase II Stratum 1: Children with LGG characterized by a BRAF truncated fusion (KIAA1549 and similar translocations)
Arm/Group | Phase II Stratum 1 | Phase II Stratum 2
Number analyzed (Participants) | 27 | 21
percentage of participants
  Progression Free Survival at 12 cycles | 59.1 [37.1 to 75.7] | 90.0 [65.6 to 97.4]
  Overall Survival at 12 cycles | 95.8 [73.9 to 99.4] | 100 [NA to NA] — All patients are surviving

ADVERSE EVENTS:
Time Frame: From time of first dose of investigational product through 30 days after last dose (maximum 96 weeks treatment duration)
Description: For non-serious adverse events, maximum AE grades 3 or 4 were reported regardless of attribution. Only one instance of each AE name is reported per subject.
Groups:
- Phase I Dose Level 2: Children with recurrent tumors signaling through the Ras/Raf pathway will be treated in 3 strata to define the activity of MEK162. S1: Children with LGG characterized by a BRAF truncated fusion (KIAA1549 and similar translocations). S2: Children with NF1 and LGG. S 3: Children with tumors involving the Ras/Raf pathway not included in strata 1 or 2.
  MEK162: • MEK162 is currently supplied as film-coated tablets in dose strength of 15 mg. The film-coated tablets consist of MEK162 drug substance, lactose monohydrate, microcrystalline cellulose, colloidal silicon dioxide, croscarmellose sodium, magnesium stearate, and a commercial film coating. The original tablets are yellow to dark yellow capsule-shaped
- Phase II Stratum 4 (Surgical Arm, Target Validation): Starting dose of 32 mg/m2/dose BID for patients who meet criteria for stratum 1, 2, or 3 for whom tumor biopsy and/or resection is clinically indicated.
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level 2 | Phase I Dose Level 3 | Phase I Dose Level 4 | Phase I Dose Level 5 | Phase II Stratum 1 | Phase II Stratum 2 | Phase II Stratum 3 | Phase II Stratum 4 (Surgical Arm, Target Validation)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 0/3 | 0/6 | 0/27 | 0/22 | 0/30 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/3 | 2/3 | 3/3 | 4/6 | 12/27 | 6/22 | 12/30 | 5/7
Other Adverse Events (participants affected / at risk) | 1/4 | 2/3 | 2/3 | 1/3 | 6/6 | 19/27 | 13/22 | 20/30 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Phase I Dose Level 1 (N=4) | Phase I Dose Level 2 (N=3) | Phase I Dose Level 3 (N=3) | Phase I Dose Level 4 (N=3) | Phase I Dose Level 5 (N=6) | Phase II Stratum 1 (N=27) | Phase II Stratum 2 (N=22) | Phase II Stratum 3 (N=30) | Phase II Stratum 4 (Surgical Arm, Target Validation) (N=7)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1/21 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1/21 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0/21 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1/21 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1/21 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0/21 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 4 | 0/21 | 1 | 0
Edema face (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0/21 | 0 | 0
Edema limbs (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1/21 | 0 | 2
Flu like symptoms (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0/21 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0/21 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 2 | 0
Bone infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0/21 | 0 | 0
Bronchial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1/21 | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1/21 | 0 | 1
Infective myositis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0/21 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0/21 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1/21 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1/21 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 2/21 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1/21 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0/21 | 0 | 0
CPK increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0/21 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1/21 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2/21 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0/21 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1/21 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0/21 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 3 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1/21 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0/21 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 2 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0/21 | 2 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0/21 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0/21 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0/21 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0/21 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0/21 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1/21 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1/21 | 0 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 0 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0/21 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 1 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Phase I Dose Level 1 (N=4) | Phase I Dose Level 2 (N=3) | Phase I Dose Level 3 (N=3) | Phase I Dose Level 4 (N=3) | Phase I Dose Level 5 (N=6) | Phase II Stratum 1 (N=27) | Phase II Stratum 2 (N=22) | Phase II Stratum 3 (N=30) | Phase II Stratum 4 (Surgical Arm, Target Validation) (N=7)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2/21 | 0 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1/21 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0/21 | 0 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0/21 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2/21 | 0 | 0
Edema limbs (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0/21 | 0 | 0
Edema trunk (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0/21 | 1 | 0
Fever (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0/21 | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 0 | 0
Irritability (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 0 | 1
Papulopustular rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1/21 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 2 | 0
Peritoneal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0/21 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0/21 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0/21 | 0 | 0
Pharyngeal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0/21 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0/21 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1/21 | 1 | 0
CPK increased (Investigations) | 1 | 1 | 0 | 0 | 2 | 3 | 5/21 | 7 | 2
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1/21 | 1 | 0
Investigations - Other, specify (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0/21 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0/21 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 1 | 0/21 | 1 | 0
Weight gain (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 1/21 | 5 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0/21 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1/21 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0/21 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1/21 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0/21 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0/21 | 2 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1/21 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1/21 | 0 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1/21 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0/21 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0/21 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1/21 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1/21 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0/21 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0/21 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0/21 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1/21 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 3/21 | 4 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 3 | 3/21 | 3 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0/21 | 1 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0/21 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2/21 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/39/NCT02285439/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT02285439/ICF_001.pdf